CLINICAL TRIAL: NCT01668888
Title: Progranulin and CTRP3 in Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: KoreaHealth_Progranulin
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Apparently Helathy Subjects

SUMMARY:
Inflammation has been known to be a pivotal pathogenic mechanism of obesity-related disorders such as type 2 diabetes, metabolic syndrome and atherosclerosis. Adipose tissue functions as a major endocrine organ by adipokine mediated modulation of a number of signaling cascades in target tissues, that has pro-inflammatory or anti-inflammatory activities. Progranulin and CTRP3 are recently discovered novel adipokines. Therefore, the investigators tried to clarify the clinical meaning of these two adipokines in the subjects with or without metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* 20<age<80
* apparently healthy subjects

Exclusion Criteria:

* a history of CVD
* diabetes
* stage 2 hypertension
* malignancy
* severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects who visited for a routine health check-up at the Health Promotion Center of Korea University Guro Hospital were enrolled using predefined inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Serum concentration of progranulin in the subjects with metabolic syndrome | 12week
Serum concentration of CTRP3 in the subjects with metabolic syndrome | 12week

SECONDARY OUTCOMES:
The relationship of serum progranulin levels with cardiovascular risk factors | 12 week
The relationship of serum CTRP3 levels with cardiovascular risk factors | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoo HJ, Hwang SY, Hong HC, Choi HY, Yang SJ, Choi DS, Baik SH, Bluher M, Youn BS, Choi KM. Implication of progranulin and C1q/TNF-related protein-3 (CTRP3) on inflammation and atherosclerosis in subjects with or without metabolic syndrome. PLoS One. 2013;8(2):e55744. doi: 10.1371/journal.pone.0055744. Epub 2013 Feb 7. PMID 23409033